CLINICAL TRIAL: NCT03328039
Title: uSing Wearable TEchnology to Predict Perioperative High-riSk Patient Outcomes
Acronym: STEPS
Status: Completed | Type: Observational
Sponsor: Cardiff University (Other)
Collaborators: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Other Study IDs: SPON1571-16
Record Dates: First submitted 2016-12-08; First posted 2017-11-01 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2018-02

CONDITIONS: Perioperative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Garmin wearable device — Physiological data capture only

SUMMARY:
This is an observational, non-interventional study to assess the equivalence of wearable monitors with formal CPET testing for the prediction of physiological reserve before major surgery.

DETAILED DESCRIPTION:
This project will exploit the rapid development of wearable technology to allow perioperative risk prediction to become logistically easier, cost effective and used more broadly. It will use low cost wearable technology to complement or act as a surrogate to complex CPET testing performed for perioperative risk stratification. The data gained from a Garmin Vivosmart HR+ wearable device, will be used in the community by patients awaiting surgery, and will be correlated with key CPET indices including anaerobic threshold and peak VO2. Ultimately, this study aims to assess whether wearable technology can provide the data needed for the formation of prediction models to risk assess perioperative outcomes in patients undergoing high-risk elective surgery. In addition, an International Physical Activity Questionnaire (IPAQ) will be completed to compare the activity captured with self-reported activity. This will be combined with frailty scores and handgrip strength as is routinely collected during CPET. Finally, a saliva based genetic analysis will be conducted on genetic variations known to be of significance in critical illness and response to physical stress. This will be delivered by a laboratory (Fitness Genes) that has developed a bespoke panel of genetic markers ideally suited to this patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older with capacity to consent
* Clinical indications for planned CPET testing before planned major elective surgery

Exclusion Criteria:

* Atrial fibrillation
* Nickel allergy
* Unable to wear a watch
* Unable to conduct CPET
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recently, low-cost, wearable activity monitors have become very popular. They can record lots of information about a person's general health and activity. In this study, we would like to see if an activity monitor can help predict a person's risk of developing complications after having major surgery.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Successful recoding of accelerometer data | 7 days
  Successful recoding of accelerometer data

CONTACTS AND LOCATIONS:
Overall Officials: Matt Morgan, PhD, Principal Investigator — Cardiff University
Locations (1):
- University Hospital of Wales, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Only on request.

REFERENCES:
- [Derived] Jones L, Tan L, Carey-Jones S, Riddell N, Davies R, Brownsdon A, Kelson M, Williams-Thomas R, Busse M, Davies MM, Morgan MPG. Can wearable technology be used to approximate cardiopulmonary exercise testing metrics? Perioper Med (Lond). 2021 Mar 16;10(1):9. doi: 10.1186/s13741-021-00180-w. PMID 33722305